CLINICAL TRIAL: NCT01409174
Title: IPI-Biochemotherapy for Chemonaive Patients With Metastatic Melanoma
Brief Title: IPI Biochemotherapy for Chemonaive Patients With Metastatic Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual, closed in Phase I.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0073; NCI-2011-02768 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Melanoma
Keywords: Melanoma; Metastatic; IPI-Biochemotherapy; Chemonaive; Advanced stage IV; Unresectable stage III melanoma; 1.0 cm or larger; Ipilimumab; Yervoy; BMS-734016; MDX010; Interferon Alpha-2b; Intron A; Temozolomide; Temodar; Cisplatin; Platinol-AQ; Platinol; CDDP; Interleukin-2; IL-2; Aldesleukin; Proleukin
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — Ipilimumab; Temozolomide; Cisplatin; Interferon alpha-2; Introns; Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ipilimumab + Chemotherapy (Experimental): Ipilimumab starting 1 mg/kg by vein (IV) Day 1 each cycle; Temozolomide 200 mg/m^2 orally Days 2-5 of Induction; Cisplatin 25 mg/m^2 IV for Days 2-4 of Induction; Interferon alfa-2b 5 million U/m2 subcutaneously on Days 1-5 of each cycle Induction + Consolidation; and Interleukin-2 9 million IU/m^2 IV as a continuous infusion on Days 2-5 of Induction + Consolidation.
  Interventions: Drug: Ipilimumab; Drug: Temozolomide; Drug: Cisplatin; Drug: Interferon Alfa-2b; Drug: Interleukin-2

INTERVENTIONS:
Drug: Ipilimumab — Phase I Starting dose: 1 mg/kg by vein over 90 minutes on Day 1 of each 3 week cycle for Induction 12 weeks, then Day 1 of Cycle 1 for Consolidation 12 weeks and Day 1 of each 12 week cycle in Maintenance.
  Phase II dose: Maximum tolerated dose (MTD) from Phase I.
  Other Names: Yervoy; BMS-734016; MDX010
Drug: Temozolomide — 200 mg/m^2 by mouth 1 time a day on Days 2-5 of each Induction cycle (four 3 week cycles).
  Other Names: Temodar
Drug: Cisplatin — 25 mg/m^2 by vein over 1 hour on Days 2-4 of each Induction cycle (four 3 week cycles).
  Other Names: Platinol-AQ; Platinol; CDDP
Drug: Interferon Alfa-2b — 5 million U/m2 subcutaneously on Days 2-6 of each 3 week Induction cycle (four 3 week cycles) and each 4 week Consolidation cycle (three 4 week cycles).
  Other Names: Intron A
Drug: Interleukin-2 — 9 million IU/m^2 by vein as a continuous infusion on Days 2-5 of each 3 week Induction cycle (four 3 week cycles) and each 4 week Consolidation cycle (three 4 week cycles).
  Other Names: IL-2; Aldesleukin; Proleukin

SUMMARY:
The goal of the Phase I part of this clinical research study is to find the highest tolerable dose of the drug Yervoy (ipilimumab) that can be given with the drugs Temodar (temozolomide), Intron-A (interferon alfa-2b), Proleukin (aldesleukin, IL-2), and Platinol (cisplatin) to patients with metastatic melanoma. The safety of this combination will also be studied in Phase I. The goal of Phase II is to learn if this combination can help to control metastatic melanoma. Note: The study was closed following Phase I enrollment.

Ipilimumab, interferon alfa-2b, and aldesleukin are designed to block the activity of cells that decrease the immune system's ability to fight cancer.

Temozolomide is designed to stop cancer cells from making new DNA (the genetic material of cells). This may stop the cancer cells from dividing into new cells.

Cisplatin is designed to poison the cancer cells, which may cause them to die.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. Up to 6 groups of 3 participants will be enrolled in the Phase I portion of the study, and up to 46 participants will be enrolled in Phase II.

***Study was halted early due to slow accrual in the Phase I portion without opening Phase II. ***

If you are enrolled in the Phase I portion, the dose of ipilimumab you receive will depend on when you joined this study. The first group of participants will receive the lowest dose level of ipilimumab. Each new group will receive a higher dose of ipilimumab than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of ipilimumab is found.

If you are enrolled in the Phase II portion, you will receive ipilimumab at the highest dose that was tolerated in the Phase I portion.

All participants will receive the same dose level of cisplatin, temozolomide, interferon alfa-2b and IL-2.

If you develop intolerable side effects while on study, your dose of IL-2 may be lowered 1-2 times until the side effects get better.

Catheter:

If you are found to be eligible to take part in this study, you will have a central venous catheter (CVC) inserted, if you do not already have one. A CVC is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form.

Study Drug Administration:

The study drugs will be given in 3 stages: induction, consolidation, and maintenance.

Induction:

Induction will last 12 weeks. You will receive the study drugs in up to four 3-week cycles:

* You will receive ipilimumab by vein over 90 minutes on Day 1 of each cycle.
* You will take temozolomide by mouth 1 time a day on Days 2-5 of each cycle. You should take temozolomide on an empty stomach at least 2 hours before or after a meal. Do not open the capsule, mix it with food, or chew it.
* You will receive cisplatin by vein over 1 hour on Days 2-4 of each cycle.
* You will receive aldesleukin by vein as a continuous infusion on Days 2-5 of each cycle.
* You will receive interferon alfa-2b as an injection under your skin on Days 2-6 of each cycle.

Consolidation:

Consolidation will last 12 weeks. You will receive the study drugs in three 4-week cycles.

* You will receive ipilimumab by vein over 90 minutes on Day 1 of consolidation.
* You will receive interferon alfa-2b as an injection under your skin on Days 1-5 of each cycle.
* You will receive aldesleukin by vein as a continuous infusion on Days 2-5 of each cycle.

Maintenance:

Maintenance will last about 1½ years. You will receive ipilimumab by vein over 90 minutes on Day 1 of up to six 12-week cycles.

Other Drugs:

You will be given other drugs to help decrease the risk of side effects. The study staff will tell you about these drugs, how they will be given, and the possible risks.

Study Visits:

Before each cycle (+/- 3 days):

* You will be asked about any drugs you may be taking and any side effects you may have had.
* Your performance status will be recorded.
* Your vital signs will be measured.
* If you are able to become pregnant, you will have a blood (about 1 teaspoon) or urine pregnancy test.

Every week, blood (about 1 teaspoon) will be drawn for routine tests. Before each cycle, some of this blood will be used to check your liver and kidney function.

At the end of each cycle, you will have a physical exam, including measurement of your weight. Any tumor that can be felt with the hands will be measured during the physical exam to see if it has changed size.

Every 2 cycles (+/- 7 days), you will have a chest x-ray and CT or MRI scans to check the status of the disease.

Anytime the doctor thinks it is needed, photos of the skin lesions will be taken. Your private areas will be covered (as much as possible), and a picture of your face will not be taken unless there are lesions on your face.

Length of Study:

You may continue taking the study drugs for up to 2 years. You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over once you have completed the end-of-treatment visit and follow-up.

End-of-Treatment Visit:

Within 14 days after you stop the study therapy, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs and weight.
* Your performance status will be recorded.
* You will be asked about any drugs you may be taking and any side effects you may have had.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* If the doctor thinks it is needed, you will have a CT or MRI scan.

Follow-Up:

Every 2 months for up to 3 years, you will be contacted by phone or during a clinic visit to see how you are doing.

This is an investigational study. Temozolomide, cisplatin, ipilimumab, interferon alfa-2b, and aldesleukin are FDA approved and commercially available to treat metastatic cancer. However, it is investigational to give temozolomide to patients with metastatic melanoma.

Up to 64 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically documented diagnosis of advanced stage IV or unresectable stage III melanoma are eligible for Phase I and Phase II
2. They must have recurrent melanoma with measurable or evaluable sites of disease, 1.0 cm or larger, in order to assess the response to treatment by the immune-related response criteria
3. Phase I: Patients with prior therapy who do not have alternative treatment of higher priority will be eligible. Phase II: patients should not have been previously treated with cytotoxic drugs or drugs included in IPI-Biochemotherapy or regional therapy for metastatic malignant melanoma. Prior adjuvant interferon is permitted. Prior adjuvant Ipilimumab therapy is not permitted. Prior therapy with targeted therapy including but not limited to B-RAF, MEK inhibitors etc. is allowed. At least three weeks should have passed since the last dose of prior adjuvant interferon therapy and prior targeted therapies and patient has fully recovered from toxicities of drugs. Prior radiation therapy for metastatic melanoma is permitted provided the patient has unirradiated metastatic sites for response evaluation and has fully recovered from its toxicity.
4. Patients between 18 years of age and 65 years of age with an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2 will be eligible.
5. They should have normal blood counts with a (white blood cell (WBC) count of more than or equal to 3000/mm^3 an absolute neutrophil count of more than or equal to 1500/mm^3 and a platelet count of more than 100,000/mm^3 and have no impairment of renal function (serum creatinine less than 1.1 mg/dl for females and less than 1.4 mg/dl for males), hepatic function (serum bilirubin level of less than 1.2 mg/dl) and no evidence of significant cardiac or pulmonary dysfunction.
6. They should have no significant intercurrent illness such as an active infection associated with fever lasting more than 24 hours requiring antibiotics, uncontrolled psychiatric illness, hypercalcemia (calcium greater than 11 mg), or active GI bleeding.
7. Females of child-bearing potential (non-childbearing is defined as greater than one year post-menopausal or surgically sterilized) must use acceptable contraceptive methods( abstinence, intrauterine device, oral contraceptive or double barrier devices) and must have a negative serum or urine pregnancy test within 72 hours prior to beginning treatment on this trial. Sexually active men must also use acceptable contraceptive methods for the duration of time on study.

Exclusion Criteria:

1. Patients with bone metastases only.
2. Patients with brain metastases unless all of their metastatic brain lesions have been resected or treated with stereotactic radiotherapy with gamma rays and they are off corticosteroids. Patient should not have significant brain edema. Patients with spinal cord compression and leptomeningeal disease are not eligible. Patients with treated central nervous system (CNS) metastases are not eligible for the neoadjuvant treatment cohort in Phase II. No major surgery or radiation therapy within 21 days before starting treatment.
3. Patients with significant cardiac illness such as symptomatic coronary artery disease or previous history of myocardial infarction, impaired left ventricle function (Ejection Fraction less than 50%) on account of any organic disease such as hypertension or valvular heart disease or serious cardiac arrhythmia requiring therapy. Patients will be evaluated by the investigator or his designee.
4. Patients with significant impairment of pulmonary function on account of chronic bronchitis or chronic obstructive pulmonary disease (COPD) which has resulted in impairment of vital capacity of forced expiratory volume at one second (FEV1) to less than 75% of predicted normal values.
5. Patients with symptomatic effusions on account of pleural, pericardial or peritoneal metastases of melanoma.
6. Patients who are unable to return for follow-up visits as required by this study.
7. Autoimmune disease: Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (eg, rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [eg, Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome and Myasthenia Gravis).
8. Patients with a history of second malignant tumor, other than the common skin cancers - basal and squamous carcinomas, within the past 3 years and uncertainty about the histological nature of the metastatic lesions. Cases with other types of malignancies should be reviewed and decided by the PI of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Tumor Response by Participant using immune-related response criteria (irRC) | End of 2 cycles, 24 weeks
  Tumor assessments using irRC modified World Health Organizations (WHO) criteria: Immune-Related Complete Response (irCR): Complete disappearance of all tumor lesions. Immune-Related Partial Response (irPR): decrease of 50% or greater. Immune-Related Progressive Disease (irPD): At least 25% increase in sum of products of all index lesions over baseline sum of products of diameters (SPD) calculated for index lesions. Assessment include photographic measurement of skin lesions, computed tomography scans and/or magnetic resonance imaging tumor assessments until documented tumor progression.

CONTACTS AND LOCATIONS:
Overall Officials: Rodabe N. Amaria, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org